CLINICAL TRIAL: NCT01085110
Title: Neurophysiological Characterization of Persistent Pain After Laparoscopic Inguinal Hernia Repair
Brief Title: Persistent Pain After Laparoscopic Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Principal Investigator, Gitte Linderoth, M.D., Rigshospitalet, Denmark
Other Study IDs: H-2-2009-126-A
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Pain, Postoperative; Neuropathic Pain; Postherniotomy Pain
Keywords: Groin hernia; Chronic pain; QST; Quantitative sensory testing; Persistent postoperative pain; Laparoscopic inguinal herniotomy; Postherniotomy Pain after laparoscopic inguinal herniotomy; laparoscopic inguinal hernia repair
MeSH Terms: conditions — Pain, Postoperative; Neuralgia; Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persistent Pain patients: Patients with persistent postherniotomy pain after laparoscopic operation and pain related impaired daily function

SUMMARY:
Describe and characterizes laparoscopic postherniotomy patients with persistent moderate/severe pain affecting every day activities - including detailed quantitative sensory assessment

ELIGIBILITY:
Inclusion Criteria:

* Male patients > 18 yrs
* No sign of hernia recurrence
* Chronic groin pain lasting more than 3 months
* Moderate/severe pain related impairment of everyday activities

Exclusion Criteria:

* Other causes of persistent pain in groin region (hip, other surgical procedures)
* Drug or alcohol abuse
* Conflicting neurological disorders

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent pain after laparoscpic inguinal hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Linderoth, MD, Principal Investigator — Section of Surgical Pathophysiology, Rigshospitalet; Henrik Kehlet, MD, Proff, Study Director — Section of Surgical Pathophysiology, Rigshospitalet
Locations (1):
- Section of Surgical Pathophysiology, Rigshospitalet, Copenhagen University, Copenhagen, Denmark